CLINICAL TRIAL: NCT07104318
Title: Randomized Clinical Trial of Personalized vs Standard of Care Treatment for Helicobacter Pylori Eradication Among Veterans: "VA Eradicate HP"
Brief Title: Personalized vs Standard of Care Treatment for Helicobacter Pylori Eradication Among Veterans
Acronym: VA EradicateHP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INFB-001-25S; H230142 (Other: VA San Diego Healthcare System IRB)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Helicobacter Pylori
Keywords: Helicobacter pylori; H. pylori; Randomized Intervention Study; CYP2C19; antibiotic susceptibility; personalized treatment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized bismuth-based quadruple therapy or clarithromycin triple therapy (Experimental): Participants allocated to the experimental group receive a personalized treatment based on clarithromycin (CLR) and amoxicillin susceptibility and CYP2C19 metabolizer profile status as follows:
  1. CLR or amoxicillin resistant/CYP2C19 normal/rapid/ultrarapid metabolizers receive bismuth quadruple therapy (BQT) with optimized PPI (bismuth 524mg QID, metronidazole 500mg QID, tetracycline 500MG QID, and omeprazole 20 mg QID) for 14 days.
  2. CLR or amoxicillin resistant/CYP2C19 intermediate/poor metabolizers receive BQT with standard PPI (BQT + omeprazole 20mg BID) for 14 days.
  3. CLR and amoxicillin susceptible/CYP2C19 normal/rapid/ultrarapid metabolizers receive CLR triple therapy with optimized PPI (amoxicillin 1000mg BID, clarithromycin 500mg BID, and omeprazole 20mg QID) for 14 days.
  4. CLR and amoxicillin susceptible/CYP2C19 intermediate/poor metabolizers receive CLR triple therapy with standard PPI (CLR triple therapy + omeprazole 20mg BID).
  Interventions: Drug: Bismuth quadruple therapy with optimized PPI; Drug: Bismuth quadruple therapy with standard PPI; Drug: Clarithromycin triple therapy with optimized PPI; Drug: Clarithromycin triple therapy with standard PPI
- Standard bismuth-based quadruple therapy (Active Comparator): Participants allocated to this group receive standard bismuth-based quadruple therapy (BQT), which is first-line treatment according to US clinical guidelines. BQT consists of bismuth subsalicylate 524mg QID (or bismuth subcitrate if salicylate allergy), tetracycline 500mg QID, metronidazole 500mg QID, and twice daily standard dose PPI (omeprazole 20mg BID) for 14 days.
  Interventions: Drug: Standard bismuth quadruple therapy

INTERVENTIONS:
Drug: Bismuth quadruple therapy with optimized PPI — Bismuth 524mg QID, Metronidazole 500mg QID, Tetracycline 500MG QID, and Omeprazole 20 mg QID for 14 days.
  Arms: Personalized bismuth-based quadruple therapy or clarithromycin triple therapy
Drug: Bismuth quadruple therapy with standard PPI — Bismuth 524mg QID, Metronidazole 500mg QID, Tetracycline 500mg QID, and Omeprazole 20mg (active BID + placebo BID) for 14 days.
  **NOTE: placebo tablets are used to maintain the same number of pills in all study arms and preserve blinding
  Arms: Personalized bismuth-based quadruple therapy or clarithromycin triple therapy
Drug: Clarithromycin triple therapy with optimized PPI — Amoxicillin 1000mg (active BID + placebo BID), Clarithromycin 500mg (active BID + placebo BID), and Omeprazole 20mg QID for 14 days. **NOTE: placebo tablets are used to maintain the same number of pills in all study arms and preserve blinding
  Arms: Personalized bismuth-based quadruple therapy or clarithromycin triple therapy
Drug: Clarithromycin triple therapy with standard PPI — Amoxicillin 1000mg (active BID + placebo BID), Clarithromycin 500mg (active BID + placebo BID), and Omeprazole 20mg (active BID + placebo BID) for 14 days. **NOTE: placebo tablets are used to maintain the same number of pills in all study arms and preserve blinding
  Arms: Personalized bismuth-based quadruple therapy or clarithromycin triple therapy
Drug: Standard bismuth quadruple therapy — Bismuth 524mg QID, Metronidazole 500mg QID, Tetracycline 500mg QID, and Omeprazole 20mg (active BID + placebo BID) for 14 days. **NOTE: placebo tablets are used to maintain the same number of pills in all study arms and preserve blinding
  Arms: Standard bismuth-based quadruple therapy

SUMMARY:
The primary objective of this study is to compare the Helicobacter pylori (H. pylori) eradication rate following empiric bismuth-based quadruple therapy (BQT) versus a personalized H. pylori treatment strategy in treatment-naïve Veterans with confirmed H. pylori infection.

This study is an eight-week, parallel two-arm, double-blinded, prospective, single-site randomized clinical trial designed to test the hypothesis that personalized H. pylori therapy achieves higher eradication rates compared to the standard empiric BQT regimen. Secondary outcomes include comparisons of treatment adherence, tolerability, and the incidence of treatment-related side effects and adverse events between the two groups. A total of 360 treatment-naïve Veterans with active H. pylori infection, confirmed by a positive H. pylori stool antigen test (HPsAg), will be enrolled, randomized, and analyzed at the VA San Diego Healthcare System (VASDHS). Participants who meet eligibility criteria and provide informed consent will be randomized in a 1:1 ratio to receive either a 14-day personalized H. pylori treatment regimen (n=180) or a standard 14-day empiric BQT regimen (n=180).

Participants randomized to personalized therapy will receive H. pylori treatment that incorporates 1) standard or optimized proton pump inhibitor (PPI) dosing according to participants' CYP2C19 metabolizer phenotype, and 2) tailored antibiotics according to participants' noninvasive (stool) H. pylori antibiotic susceptibility testing (AST). All participants will complete a baseline questionnaire and provide pre-treatment stool and blood samples for H. pylori AST and serum CYP2C19 testing, respectively. Follow-up will include brief telephone interviews during week 1 and week 2 of treatment and again two weeks post-treatment to assess adherence and monitor for adverse events. Cure will be assessed using a post-treatment stool antigen test (HPsAg) at week 8 (four weeks after completing therapy).

ELIGIBILITY:
Inclusion Criteria:

* Adult Veterans ages 18 years or older, irrespective of sex/gender (male, female, non-binary, other preferred classification).
* Treatment-naïve patients with active H. pylori infection as determined by a positive H. pylori stool antigen (HPsAg), gastric biopsy, or urease breath test. All individuals who test positive based on a non-HPsAg modality will need to have a positive HPsAg documented within 4 weeks of enrollment to be considered eligible.
* Subjects who can understand and sign written informed consent.

Exclusion Criteria:

The investigators will exclude individuals with:

* Severe gastrointestinal (GI) symptoms that limit the ability to tolerate study medications. Note: The presence of symptoms or GI diagnoses such as irritable bowel syndrome or gastroesophageal reflux does not impact H. pylori eradication and will not be exclusion criteria unless deemed that symptom severity will impact adherence.
* Conditions where urgent H. pylori treatment is recommended (i.e., active peptic ulcer disease (PUD) complicated by bleeding, perforation, or obstruction; gastric neoplasia including MALT lymphoma). Active PUD is defined as having a gastric or duodenal ulcer confirmed on an upper endoscopic procedure in the 4 weeks prior to eligibility determination.
* Inability to be safely off of PPI for two weeks to allow for accurate post-treatment HPsAg testing. These conditions include Barrett's esophagus with dysplasia, active PUD, severe esophagitis defined as Los Angeles Classification C or D esophagitis.
* Allergy or severe intolerance/contraindication to any of the treatment components. Note: In patients with penicillin allergy, metronidazole is often substituted for amoxicillin in PPI clarithromycin triple therapy. However, this alternative regimen demonstrates higher failure rates vs. PPI-clarithromycin triple therapy with amoxicillin among Veterans and thus the investigators elected to exclude patients with penicillin allergy.
* Severe medical comorbidity that is a threat to life. This includes, but is not limited to, coronary artery disease with myocardial infarction or equivalent (e.g., cerebrovascular event) within 12 months, unstable angina or congestive heart failure, cardiac or vascular stent placement within 12 months, chronic obstructive pulmonary disease requiring home oxygen, decompensated cirrhosis, end-stage renal disease, other diseases that limit life expectancy to less than 5 years.
* Any prior history of upper gastrointestinal surgery or gastric cancer diagnosis.
* Past liver transplant or allogenic bone marrow transplant, given that pharmacogenomic testing is inaccurate for these patients.
* Any history of recurrent Clostridioides difficile infection (CDI), defined as an episode of CDI occurring within 8 weeks of a previous CDI episode; or any episode of CDI within the preceding 12 months.
* Evidence of any overt gastrointestinal bleeding.
* History of photosensitive reactions to any medications.
* Women who are pregnant, lactating, or of childbearing age without reliable contraception (Note: all women of childbearing age will be asked to submit a urine pregnancy test prior to enrollment).
* Prior CYP2C19 or PHASER testing or HP antimicrobial susceptibility profiling before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication success | 4-6 weeks after treatment
  The primary outcome is H. pylori eradication success, defined as negative post-treatment H. pylori stool antigen (HPsAg) testing. Post-treatment persistent positive HPsAg indicates eradication treatment failure; equivocal tests will be conservatively counted as a treatment failure, along with participants who fail to complete follow up testing within the prespecified timeframe (intention-to-treat analysis). All participants must be off proton pump inhibitors (PPIs) for a minimum of 2 weeks, and off antibiotics or bismuth for at least 4 weeks prior to HPsAg testing. HPsAg testing will be performed between 4-6 weeks post-treatment.

SECONDARY OUTCOMES:
Treatment adherence | Weeks 1 and 2 after treatment initiation
  Patient-reported treatment adherence will be evaluated using the validated Adherence to Refills and Medications Scale (ARMS) and pill counts obtained during telephone interviews conducted in weeks 1 and 2 following treatment initiation. Adherence will be defined as >90% of the treatment regimen consumed.
Treatment-emergent side effects/adverse events | Weeks 1 and 2 after treatment initiation, 6 weeks after treatment completion
  Participant-reported side effects and adverse events will be collected during telephone interviews conducted in weeks 1 and 2 following treatment initiation, and in week 6 following treatment completion. Treatment-emergent adverse events will be classified using the Medical Dictionary for Regulatory Activities terminology (MedDRA).

CONTACTS AND LOCATIONS:
Overall Officials: Shailja Shah, MD MPH, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No